CLINICAL TRIAL: NCT02401828
Title: The Dolutegravir Antiretroviral Mono-Therapy for HIV Trial
Acronym: DOMONO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Bart Rijnders, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL51858.078.14
Record Dates: First submitted 2015-03-19; First posted 2015-03-30 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - Direct Switch (Experimental): Direct switch from cART to Dolutegravir mono-therapy at baseline. Dolutegravir single tablet 50mg QD, once a day. Duration = 48 weeks
  Interventions: Drug: Dolutegravir
- Group B - Delayed Switch (Experimental): Delayed switch from cART to Dolutegravir mono-therapy at week 24 from baseline. Dolutegravir single tablet 50mg QD, once a day. Duration = 48 weeks
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — Switch from combination antiretroviral therapy to dolutegravir monotherapy
  Other Names: Tivicay; S/GSK1349572

SUMMARY:
48-week open label randomized phase IV investigator initiated intervention study. The purpose of this study is to evaluate whether HIV-1 suppression can be maintained by DTG monotherapy in HIV-1 infected, virologically suppressed patients on cART.

104 adults fulfilling the in and exclusion criteria and on stable cART will be randomized over 2 investigational arms.

The first arm will contain the direct switch population. This population will switch directly from stable cART to Dolutegravir mono-therapy on baseline visit.

The second arm will contain the delayed-switch population. This group will switch from stable cART to Dolutegravir monotherapy 24 weeks after baseline visit.

The main goal is to investigate if Dolutegravir mono-therapy could be non-inferior to cART in virological suppressed HIV-1 infected adults.

If a interim analysis (performed when 40 patients on dolutegravir monotherapy have passed week 12) shows that it is safe to continue the study, an additional 30 patients will be included on top of the 104 patients needed for the primary endpoint analysis. In contrast to the primary endpoint population, these additional 30 patients will have a CD4 nadir <200 but a CD4 >350 at the time of the screening visit. Besides that, these 30 patients will have to fulfill all other in and exclusion criteria of the primary endpoint population (specifically a viral load never >100.000). These 30 patients are part of a pilot study looking at the possibility to broaden the eligible population in a future larger randomized clinical trial.

DETAILED DESCRIPTION:
DTG Monotherapy will be considered non-inferior to cART if the lower bound of the one sided 97.5%CI for the difference in proportion of patients reaching the primary endpoint is not lower than -12%. For this purpose, a sample size of 52 per arm would provide 80% power at alpha 0.025 to establish non-inferiority of DTG monotherapy compared with cART when the primary endpoint success rate is 95% in both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 positive by ELISA or Western Blot or Plasma HIV-RNA >1000 c/ml.
* 18 years or older.
* HIV-RNA ≤50 copies/mL for ≥24 weeks.
* Historical baseline HIV-RNA plasma load <100.000 c/ml
* CD4 count nadir pre-cART ≥200 cells/mm3
* Not on strong UGT1A1 or CYP3A4 inducing agents as stated in DTG SPC.
* General medical condition does not interfere with trial procedures (on investigators' discretion)
* Females should have no plans of becoming pregnant during the next 18 months after the baseline visit
* Females are eligible if:

  1. They do not plan to become pregnant during the study
  2. Negative screening pregnancy test and uses one of the following methods: 1.Abstinence from penile/vaginal intercourse during the study; 2.Double barrier contraceptive methods 1 of which must be condom.

Exclusion Criteria:

* Previous virological failure on any ART.
* Patient without documented anti-HBs antibodies.
* Subjects positive for hepatitis B at screening (HBsAg+).
* Any documented genotypic HIV-1 resistance with at least low-level resistance according to stanford HIV drug resistance database
* No record of the historical baseline plasma viral load available
* Subjects with concomitant CDC-C opportunistic infections within 90 days of screening.
* Subjects with history of allergy to INI.
* Subjects with creatinine clearance <50mL/min according to CKD-EPI.
* Subjects with hepatic impairment of at least Child-Pugh B.
* Exposure to experimental drug or experimental HIV-1 vaccine within 90 days of start of DTG.
* Screening ALT >5x ULN or ALT>3xULN and bilirubin >2 ULN.
* Patient (man or woman) planning or hoping to conceive a child/become pregnant during the study
* Patients who cannot take DTG 2 hours before or 6 hours after antacids, calciumcarbonate or iron supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of dolutegravir monotherapy in maintaining virological suppression in the on-treatment population | 24 weeks
  HIV-RNA <200c/ml at week 24 after baseline

SECONDARY OUTCOMES:
Time to loss of virological response (TLOVR) in the OT population | 1 week
  Time to first of two confirmed HIV-RNA >50c/ml at least 1 week apart
Efficacy of dolutegravir monotherapy in maintaining virological suppression in the entire study population (ITT) | 24 weeks
  HIV-RNA <200c/ml at week 24 after baseline
Efficacy of dolutegravir monotherapy in maintaining virological suppression in the on-treatment population | 48 weeks
  HIV-RNA <50 & <200 at week 24 & 48
Evaluate safety of Dolutegravir monotherapy (Acquired resistance & Adverse Events according to CDC 4.0) | 60 weeks
  Acquired resistance & Adverse Events according to CDC 4.0
Evaluate the evolution of CD4 associated HIV-1 reservoir | 48 weeks
  Total/integrated HIV-DNA & 2LTR
Evaluate the number and type of INI resistance mutation in patients with virological failure | 48 weeks
  Virological failure: HIV-RNA >200c/ml
Evaluate CD4 cell count change | 48 weeks
  Compare baseline vs. 48 weeks after baseline
Evaluate changes in renal function after 24 and 48 weeks of dolutegravir monotherapy | 48 weeks
Cost effectiveness of DTG monotherapy | 48 weeks
  Cost per QALY during DTG monotherapy in comparison with the costs of therapy with the patient's own cART regimen used before study inclusion
Evaluate change in BMD after 24 and 48 weeks of dolutegravir mono-therapy | 48 weeks
Exploratory analysis of blood pressure, weight, BMI, fasting serum lipids, Framingham risk score, ATP-III treatment goals and inflammatory markers after 24wks of dolutegravir mono-therapy | 48 weeks
Efficacy of dolutegravir monotherapy in maintaining virological suppression in the on-treatment population | 12 weeks
  HIV-RNA <200c/ml and <50 at week 12 after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bart Rijnders, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Wijting IEA, Lungu C, Rijnders BJA, van der Ende ME, Pham HT, Mesplede T, Pas SD, Voermans JJC, Schuurman R, van de Vijver DAMC, Boers PHM, Gruters RA, Boucher CAB, van Kampen JJA. HIV-1 Resistance Dynamics in Patients With Virologic Failure to Dolutegravir Maintenance Monotherapy. J Infect Dis. 2018 Jul 24;218(5):688-697. doi: 10.1093/infdis/jiy176. PMID 29617822
- [Derived] Wijting I, Rokx C, Boucher C, van Kampen J, Pas S, de Vries-Sluijs T, Schurink C, Bax H, Derksen M, Andrinopoulou ER, van der Ende M, van Gorp E, Nouwen J, Verbon A, Bierman W, Rijnders B. Dolutegravir as maintenance monotherapy for HIV (DOMONO): a phase 2, randomised non-inferiority trial. Lancet HIV. 2017 Dec;4(12):e547-e554. doi: 10.1016/S2352-3018(17)30152-2. Epub 2017 Oct 26. PMID 29107562